CLINICAL TRIAL: NCT06604351
Title: The Efficacy and Safety of Bronchoscopic Cryoablation Combined With Sintilimab Plus Platinum-based Chemotherapy as First-line Treatment for Locally Advanced or Metastatic NSCLC With Central Airway Obstruction: A Phase II Study
Brief Title: Bronchoscopic Cryoablation Combined With Chemo-Immunotherapy in NSCLC With Central Airway Obstruction
Acronym: Example
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hunan Province Tumor Hospital (Other)
Responsible Party: Principal Investigator, Yongchang Zhang, Head of Medical Oncology, Director of Early Clinical Trial Center, Hunan Province Tumor Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20240827
Record Dates: First submitted 2024-08-27; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — sintilimab; 130-nm albumin-bound paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- group 1 (Experimental): Bronchial endoscopic cryoablation
  Interventions: Drug: Sintilimab, Nab-Paclitaxel, and Carboplatin

INTERVENTIONS:
Drug: Sintilimab, Nab-Paclitaxel, and Carboplatin — Cryoablation received at least 2 or more depending on the mass, with 2-3 cycles；Sintilimab 200 mg Q3W plus Nab-Paclitaxel 260mg / m2(Day 1) Q3W + carboplatin AUC 4.25 or 5 (Day 1) Q3W, 4 cycles，until 24 months

SUMMARY:
This study aimed to evaluate the efficacy and safety of bronchoscopic cryoablation combined with sintilimab plus platinum-based chemotherapy as First-line Treatment for locally advanced or metastatic NSCLC with central airway obstruction.

DETAILED DESCRIPTION:
This is a prospective interventional clinical study to evaluate the efficacy and safety of bronchoscopic cryoablation combined with sintilimab plus platinum-based chemotherapy as First-line Treatment for locally advanced or metastatic Non-small Cell Lung Cancer with central airway obstruction.

Approximately 39 patients with locally advanced or metastatic NSCLC and central airway obstruction, without EGFR-sensitive mutations (19del, L858R, and T790M), were enrolled and treated with bronchoscopic cryoablation combined with Sintilimab, Nab-Paclitaxel, and Carboplatin until disease progression, intolerable toxicity, or meeting the criteria for discontinuation of the trial drug.

The primary endpoint is the investigator-assessed objective response rate (ORR) of airway tumors. Secondary endpoints include the pathological response rate (PRR) of airway tumors, disease control rate (DCR), improvement rate of FEV1, duration of response (DOR) for airway tumors, progression-free survival (PFS), overall survival (OS), quality of life assessment, and safety. Recruitment for the study is expected to begin in mainland China around October 2024, with the trial anticipated to conclude in October 2027.

ELIGIBILITY:
Inclusion Criteria:

* Understand the requirements and contents of the clinical trial and provide a signed and dated informed consent form.
* Age≥18 years and≤80 years.
* Histologically or cytologically confirmed and documented locally advanced or metastatic non-small cell lung cancer (NSCLC) without prior systemic therapy and EGFR-sensitive mutations (19del, L858R and T790M).
* Presence of a palliative treatment lesion in the central airway that is amenable to ablation, endoscopically assessed to be≥1/3 obstruction, such as primary or metastatic malignancy to the trachea, main bronchi, intermediate bronchi, or segmental bronchi. corresponding respiratory symptoms or obstructive pneumonia is permission to be included.
* Eastern Cooperative Oncology Group (ECOG) ： 0-2.
* Predicted survival ≥ 12 weeks.
* Adequate bone marrow hematopoiesis and organ function (cardiac function, hepatic, and renal function).
* Presence of measurable lesions according to RECIST 1.1 criteria.
* Subjects with stable brain metastases may be included in the study.

Exclusion Criteria:

* Histological diagnosis of small cell, large cell lung cancer; mixed tumors will be classified based on the primary cell type; if the primary component is small cell, large cell, or neuroendocrine carcinoma, the subject will not be eligible for enrollment; however, mixed adenocarcinoma-squamous cell carcinoma is acceptable. Subjects with driver gene mutations are generally not eligible for enrollment.
* Malignant central airway obstruction with acute dyspnea or severe life-threatening symptoms of malignant airway stenosis, or assessed by the investigator to be unable to tolerate subsequent treatment; extrinsic airway compression; large pleural effusion, severe coughing, massive hemoptysis, dyspnea, or inability to cooperate; severely impaired lung function with a maximal voluntary ventilation (MVV) < 39% or inability to ambulate.
* Prior systemic therapy for locally or metastatic disease.
* Uncorrectable coagulation disorders, severe bleeding tendencies, platelet count < 50 *10^9/L, or severe coagulation dysfunction.
* Presence of symptomatic brain metastases.
* Known severe hypersensitivity to anti-PD-1 monoclonal antibodies or similar drugs (allergic reactions with CTCAE≥ grade 3 toxicity).
* Subjects with persistent or active infection, including but not limited to hepatitis B virus (HBV), hepatitis C virus (HCV), human immunodeficiency virus (HIV).
* Any concurrent malignancy other than basal cell carcinoma or cervical carcinoma in situ. (Patients with a history of malignant tumors but with no evidence of disease for≥ 3 years may be included ).
* Women who are breastfeeding or pregnant.
* Other conditions assessed by the investigator to be unsuitable for participation in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2024-09-15 (Estimated); Primary Completion 2027-10-31 (Estimated); Study Completion 2029-05-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate of Airway Tumor | Time from first dose to last dose, or up to 24 month
  The ORR for Objective response of airway tumors after cryoablation combined with immunochemotherapy was evaluated according to the investigator's Solid Tumor Response Assessment Criteria (RECIST) version 1.1, defined as the proportion of subjects who were evaluated for complete response (CR) + partial response (PR) to airway tumors after the first documented treatment

SECONDARY OUTCOMES:
Pathological Response Rate of Airway Obstruction | Time from first dose to last dose, or up to 24 month
  The pathologic response rate of airway tumors obstruction in patients treated with cryoablation combined with immunochemotherapy was evaluated according to the investigator which was defined as the proportion of subjects with endoscopically assessed airway pathologic residual tumors ≤10% after treatment recorded for the first or last time after cryoablation
Airway Obstruction Response Control Rate | Time from first subject dose to study completion, or up to 36 month
  The DCR for airway tumors obstruction in patients treated with cryoablation combined with immunochemotherapy was assessed according to the investigator's RECIST 1.1, defined as the proportion of subjects evaluated for complete (CR) + partial response (PR) and stable SD for intraairway tumors after the first recorded treatment
FEV1R improvement rate of airway obstruction | Time from first subject dose to study completion, or up to 36 month
  Calculated according to the subjects' pulmonary function measures assessed by the investigator: FEV1 (post-treatment) -FEV1 (pre-treatment)/FEV1 (pre-treatment) *100%
Airway Obstruction Response Duration | Time from first subject dose to study completion, or up to 36 month
  The duration of response in subjects with CR or PR was assessed according to the Solid Tumor Response Assessment Criteria (RECIST) version 1.1 developed by the investigators, defined as the time from the first recorded evaluated airway tumor CR or PR to airway disease progression or death
Progression-free survival | Time from first subject dose to study completion, or up to 36 month
  Progression-free survival of patients treated with cryoablation plus immunochemotherapy was assessed according to the Investigator Response Evaluation criteria (RECIST) version 1.1, defined as the duration of first documented disease progression or death from any cause
Overall survival | Time from first subject dose to study completion, or up to 36 month
  To assess overall survival, it was defined as the first dose at which the subject died from any cause
Adverse events | Time from first subject dose to study completion, or up to 36 month
  Number of participants with adverse events (AEs) according to CTCAE 5.0
Life quality score | Time from first subject dose to study completion, or up to 36 month
  Score according to EORTC QLQ-L30+QLQ-LC13 table

CONTACTS AND LOCATIONS:
Locations (1):
- Hunan Cancer hospital, Changsha, Hunan, China